CLINICAL TRIAL: NCT07146841
Title: Evaluating Cochlear Insertion Trauma and Hearing Preservation After Cochlear Implantation (CIPRES): a Study Protocol for a Randomized Single-blind Controlled Trial
Brief Title: Hearing Preservation in Cochlear Implantation Surgery
Acronym: CIPRES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Prof Dr HGXM Thomeer MD PhD, MD PhD, UMC Utrecht
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NL71233.041.19; NL8586 (Other: Netherlands Trial Register (NTR))
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sensorineural Hearing Loss
Keywords: Sensorineural Hearing Loss; Cochlear Implantation; Residual Hearing Preservation; Electrocochleography
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind trial consisting of four groups: I: RW and LW, II: RW and PM, III: CO and LW and IV: CO and PM.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1: RW and LW (Other): Combination of round window insertion and lateral wall electrode array
  Interventions: Procedure: Round window insertion; Device: Lateral wall array
- Group 2: RW and PM (Other): Combination of round window insertion and perimodiolar electrode array
  Interventions: Procedure: Round window insertion; Device: Periomodiolar electrode array
- Group 3: CO and LW (Other): Combination of cochleostomie insertion and lateral wall electrode array
  Interventions: Procedure: Cochleostomy insertion; Device: Lateral wall array
- Group 4: CO + PM (Other): Combination of cochleostomy insertion and perimodiolar electrode array
  Interventions: Procedure: Cochleostomy insertion; Device: Periomodiolar electrode array

INTERVENTIONS:
Procedure: Round window insertion — Insertion of the electrode array via the round window.
  Other Names: Round window
  Arms: Group 1: RW and LW; Group 2: RW and PM
Procedure: Cochleostomy insertion — Insertion of the electrode array via cochleostomy.
  Other Names: cochleostomy
  Arms: Group 3: CO and LW; Group 4: CO + PM
Device: Lateral wall array — Lateral wall electrode array from Advanced Bionics.
  Arms: Group 1: RW and LW; Group 3: CO and LW
Device: Periomodiolar electrode array — Perimodiolar MidScala electrode array from Advanced Bionics.
  Other Names: Perimodiolar array
  Arms: Group 2: RW and PM; Group 4: CO + PM

SUMMARY:
In order to preserve the residual hearing in patients with sensorineural hearing loss (SNHL) receiving a cochlear implant (CI), the insertion trauma to the delicate and microscopic structures of the cochlea needs to be minimized. The surgical procedure starts with the conventional mastoidectomy-posterior tympanotomy (MPT) approach to the middle ear, and is followed by accessing the cochlea, with either a cochleostomy (CO) or via the round window (RW). Both techniques have their benefits and disadvantages. Another aspect is the design of the electrode array. There are fundamentally two different designs: a *straight* lateral wall lying electrode array (LW), or a *pre-curved* perimodiolar cochlear lying electrode array (PM). Interestingly, until now, the best surgical approach and type of implant is unknown. Our hypothesis is that the combination of a RW approach and a LW lying electrode array minimizes insertion trauma, leading to better hearing outcome for SNHL patients.

ELIGIBILITY:
Inclusion Criteria:

* Severe hearing loss, CI candidate
* 18 years of age or older
* normal function of middle ear (i.e. no acute middle ear infections)
* dutch language proficiency
* choice for Advanced Bionics implant

Exclusion Criteria:

* prior otologic surgery in the implanted ear (excluding tympanostomy tube placement)
* inner ear malformation present in the ear to be implanted (i.e. ossification, Mondini malformation)
* retrocochlear pathology present in the auditory system to be implanted
* neurocognitive disorders
* sudden deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Hearing preservation | 12 months
  Hearing preservation is the main outcome, which will be expressed in percentage. Hearing preservation is calculated by using the preoperative and postoperative puretoneaudiometry (PTA).

SECONDARY OUTCOMES:
Scalar position of the electrode array | 12 months
  Scalar position of the electrode array (scala tympani or scala vestibuli assessed by CB-CT)
Electrocochleography | 12 months
  ECochG (among others amplitude in µV) and eCAP (among others amplitude in µV) potentials
Speech perception | 12 months
  Speech perception test with/without noise in CVC words correct score (in percentage) with signal to noise ratio of 10 dB.

CONTACTS AND LOCATIONS:
Overall Officials: Hans GXM Thomeer, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Rask-Andersen H, Erixon E, Kinnefors A, Lowenheim H, Schrott-Fischer A, Liu W. Anatomy of the human cochlea--implications for cochlear implantation. Cochlear Implants Int. 2011 May;12 Suppl 1:S8-13. doi: 10.1179/146701011X13001035752174. PMID 21756464
- [Background] Escude B, James C, Deguine O, Cochard N, Eter E, Fraysse B. The size of the cochlea and predictions of insertion depth angles for cochlear implant electrodes. Audiol Neurootol. 2006;11 Suppl 1:27-33. doi: 10.1159/000095611. Epub 2006 Oct 6. PMID 17063008
- [Background] Avci E, Nauwelaers T, Hamacher V, Kral A. Three-Dimensional Force Profile During Cochlear Implantation Depends on Individual Geometry and Insertion Trauma. Ear Hear. 2017 May/Jun;38(3):e168-e179. doi: 10.1097/AUD.0000000000000394. PMID 28045786
- [Background] Snels C, IntHout J, Mylanus E, Huinck W, Dhooge I. Hearing Preservation in Cochlear Implant Surgery: A Meta-Analysis. Otol Neurotol. 2019 Feb;40(2):145-153. doi: 10.1097/MAO.0000000000002083. PMID 30624395
- [Background] Fan X, Xia M, Wang Z, Zhang H, Liu C, Wang N, Hou L, Li C, Xu A. Comparison of electrode position between round window and cochleostomy inserting approaches among young children: a cone-beam computed tomography study. Acta Otolaryngol. 2018 Sep;138(9):815-821. doi: 10.1080/00016489.2018.1478127. Epub 2018 Jun 23. PMID 29936898
- [Background] Wanna GB, Noble JH, Gifford RH, Dietrich MS, Sweeney AD, Zhang D, Dawant BM, Rivas A, Labadie RF. Impact of Intrascalar Electrode Location, Electrode Type, and Angular Insertion Depth on Residual Hearing in Cochlear Implant Patients: Preliminary Results. Otol Neurotol. 2015 Sep;36(8):1343-8. doi: 10.1097/MAO.0000000000000829. PMID 26176556
- [Background] Wanna GB, Noble JH, Carlson ML, Gifford RH, Dietrich MS, Haynes DS, Dawant BM, Labadie RF. Impact of electrode design and surgical approach on scalar location and cochlear implant outcomes. Laryngoscope. 2014 Nov;124 Suppl 6(0 6):S1-7. doi: 10.1002/lary.24728. Epub 2014 May 30. PMID 24764083
- [Background] Havenith S, Lammers MJ, Tange RA, Trabalzini F, della Volpe A, van der Heijden GJ, Grolman W. Hearing preservation surgery: cochleostomy or round window approach? A systematic review. Otol Neurotol. 2013 Jun;34(4):667-74. doi: 10.1097/MAO.0b013e318288643e. PMID 23640087
- [Background] Gfeller KE, Olszewski C, Turner C, Gantz B, Oleson J. Music perception with cochlear implants and residual hearing. Audiol Neurootol. 2006;11 Suppl 1:12-5. doi: 10.1159/000095608. Epub 2006 Oct 6. PMID 17063005
- [Background] Buechner A, Brendel M, Krueger B, Frohne-Buchner C, Nogueira W, Edler B, Lenarz T. Current steering and results from novel speech coding strategies. Otol Neurotol. 2008 Feb;29(2):203-7. doi: 10.1097/mao.0b013e318163746. PMID 18223448
- [Background] Gifford RH, Dorman MF, Skarzynski H, Lorens A, Polak M, Driscoll CL, Roland P, Buchman CA. Cochlear implantation with hearing preservation yields significant benefit for speech recognition in complex listening environments. Ear Hear. 2013 Jul-Aug;34(4):413-25. doi: 10.1097/AUD.0b013e31827e8163. PMID 23446225
- [Background] Skarzynski H, Lorens A, Matusiak M, Porowski M, Skarzynski PH, James CJ. Cochlear implantation with the nucleus slim straight electrode in subjects with residual low-frequency hearing. Ear Hear. 2014 Mar-Apr;35(2):e33-43. doi: 10.1097/01.aud.0000444781.15858.f1. PMID 24556970
- [Background] Eshraghi AA, Nazarian R, Telischi FF, Rajguru SM, Truy E, Gupta C. The cochlear implant: historical aspects and future prospects. Anat Rec (Hoboken). 2012 Nov;295(11):1967-80. doi: 10.1002/ar.22580. Epub 2012 Oct 8. PMID 23044644
- [Background] Jwair S, Boerboom RA, Versnel H, Stokroos RJ, Thomeer HGXM. Evaluating cochlear insertion trauma and hearing preservation after cochlear implantation (CIPRES): a study protocol for a randomized single-blind controlled trial. Trials. 2021 Dec 9;22(1):895. doi: 10.1186/s13063-021-05878-2. PMID 34886884

DOCUMENTS (1):
  • Study Protocol (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/41/NCT07146841/Prot_000.pdf